CLINICAL TRIAL: NCT00785434
Title: Phase IV Pilot Study to Examine the Efficacy and Safety of Escitalopram in Doses up to 50 mg for the Treatment of Patients With Major Depressive Disorder (MDD).
Brief Title: Efficacy and Safety of Escitalopram Doses up to 50mg in Treatment of MDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Community Pharmacology Services Ltd (Other)
Responsible Party: Dr AG Wade, Director, CPS Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPS/04/2008
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Major Depressive Disorder
Keywords: MDD; escitalopram
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): Active escitalopram
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — Dose ranging up to 50mg

SUMMARY:
This will be an open label study of escitalopram. Patients not responsive to citalopram will be switched directly to escitalopram.

Patients will receive escalating doses of escitalopram up to a maximum of 50 mg until they either achieve remission (MADRS <9) or fail to tolerate the dose.

DETAILED DESCRIPTION:
Patients will receive escalating doses of escitalopram up to a maximum of 50 mg until they either achieve remission (MADRS <9) or fail to tolerate the dose.

Visit 1 - (Initial visit) - escitalopram 10 mg Visit 2 - (Week 2) - escitalopram 20 mg Visit 3 - (Week 4) - review visit Visit 4 - (Week 6) - MADRS <12 - continue 20 mg MADRS >12 - escitalopram 30 mg Visit 5 - (Week 8) - MADRS <8 - continue current dose MADRS >8 - escalate dose (20 mg to 30 mg or 30 mg to 35mg)

Thereafter, Patients who have achieved remission will be maintained on the remission dosage and reviewed at four weekly intervals. At any subsequent visit where the MADRS is >8 they will have a dosage increase

Patients who have not achieved remission will have dosage escalated by 5 mg at two weekly intervals until remission, a maximum dose of 50 mg is achieved or the dosage is intolerable when they will be reduced to the previous tolerable dose.

Patients will be followed up until eight months from their initial visit.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent will be obtained from each patient
* aged 18 to 65 inc
* suffering from MDD as defined by DSM IV
* have been taking citalopram in a dose of at least 20mg for at least six weeks
* an inadequate response -- defined as failure to achieve a MADRS score of <12

Exclusion Criteria:

* Significant other psychiatric disorder which would interfere with trial assessments. Co-morbid generalized anxiety disorder (GAD) and panic will be permitted where MDD is considered the primary diagnosis .
* history of mania or bipolar disorder
* Known contraindication for the use of citalopram or escitalopram.
* Significant bleeding disorder
* Prominent suicidal ideation (score more than 4 in the MADRS "suicidal thoughts" item)
* Alcohol or substance dependence in the past 6 months
* Major physical illness
* Significant liver or renal function abnormality
* Significant ECG abnormalities
* Pregnant or lactating females
* Inadequate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The number of patients achieving remission (MADRS<9). | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan G Wade, MBChB, Principal Investigator — CPS Research
Locations (1):
- CPS Research, Glasgow, United Kingdom

REFERENCES:
- [Derived] Wade AG, Crawford GM, Yellowlees A. Efficacy, safety and tolerability of escitalopram in doses up to 50 mg in Major Depressive Disorder (MDD): an open-label, pilot study. BMC Psychiatry. 2011 Mar 16;11:42. doi: 10.1186/1471-244X-11-42. PMID 21410960